CLINICAL TRIAL: NCT07407647
Title: Vaginal DHEA for Women With Gynecologic and Gastrointestinal Cancer After Radiation
Brief Title: Vaginal DHEA to Improve Vaginal Health After Radiation for Women With Gynecologic, Anal or Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Allison Quick, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-25055; NCI-2026-00035 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2026-01-14; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Anal Carcinoma; Cervical Carcinoma; Malignant Female Reproductive System Neoplasm; Rectal Carcinoma; Vaginal Carcinoma; Vulvar Carcinoma
MeSH Terms: conditions — Anus Neoplasms; Uterine Cervical Neoplasms; Rectal Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms | interventions — Specimen Handling; Dehydroepiandrosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (DHEA) (Experimental): Patients receive DHEA vaginally QD for 3 months in the absence of disease progression or unacceptable toxicity. Patients undergo vaginal swab sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Prasterone; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo vaginal swab sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Prasterone — Given vaginally
  Other Names: 17-Hormoforin; Dehydroepiandrosterone; Dehydroisoandrosterone; DHEA; Diandron; Fidelin; GL701; Therapeutic Dehydroepiandrosterone
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase II trial tests the feasibility and side effects of vaginal DHEA to improve vaginal health after radiation for women with gynecologic, anal or rectal cancer. Treatment of cancers with radiation to the abdomen can influence the vaginal microbiome (any bacteria, virus, or other organisms found in the vagina). Both menopause and radiation cause a decrease in lubrication and elasticity of the vagina and symptoms including vaginal dryness, vaginal burning and itching, vaginal bleeding, pain or burning during urination, and pain during sexual intercourse. DHEA is a type of hormone replacement therapy. It is use to improve symptoms in women during menopause and may be effective in treating these symptoms for women who have received radiation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility and tolerability of dehydroepiandrosterone (DHEA) in the post radiation setting for women with gynecologic and gastrointestinal cancers.

SECONDARY OBJECTIVES:

I. To identify changes from baseline to post-radiation in the vaginal microbiome in women with gynecologic and gastrointestinal cancers receiving vaginal DHEA.

II. To identify those who may respond to vaginal DHEA based on their pretreatment microbiome.

III. To correlate changes in vaginal exam findings, sexual function, and quality of life with changes in the vaginal microbiome.

OUTLINE:

Patients receive DHEA vaginally once daily (OD) for 3 months in the absence of disease progression or unacceptable toxicity. Patients undergo vaginal swab sample collection throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with anal, rectal, cervical, vaginal, or vulvar cancer receiving external beam radiation alone, or both external beam radiation and brachytherapy with curative intent (Participants will be consented and enrolled prior to starting treatment but will not receive intervention till after treatment is completed)
* Concurrent or prior chemotherapy is allowed
* Any prior gynecologic surgery is permitted
* Rectal surgery, including lower anterior resection and abdominoperineal resection, is permitted
* Subject must be menopausal, which is defined as age > 50 with no menses for 12 months or bilateral oophorectomy

Exclusion Criteria:

* Patients with scleroderma, mixed connective tissue disorder, and lupus will be excluded
* Patients who have received prior pelvic radiation
* Undiagnosed abnormal genital bleeding (unrelated to current diagnosis or treatment related toxicity)
* Endometrial cancer or endometrial hyperplasia
* Use of estrogen alone injectable or progestin implant therapy with 3 months before study entry
* Use of estrogen pellet or progestin injectable drug within 6 months before study entry
* Use of oral estrogen, progestin, or DHEA or intrauterine progestin within 8 weeks before study entry
* Use of vaginal estrogen (rings, creams, tablets, or gels), transdermal estrogen +/- progestin, vaginal hyaluronic acid, or pro-estrogenic herbal treatments such as black cohosh in the 4 weeks before study entry. Intravaginal moisturizers and lubricants prior to enrollment are permitted
* History of breast cancer
* Patients receiving palliative radiation therapy
* Patients who do not meet criteria for menopause

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 2 or higher adverse events | From start of treatment to 12 weeks
  Will consider this study feasible if 80% of participants are able to complete 12 weeks of dehydroepiandrosterone (DHEA) without grade 2 or higher adverse events other than vaginal discharge or due to vaginal discharge that is felt to be too bothersome to the participant.

SECONDARY OUTCOMES:
Change in vaginal microbiome | From baseline to 12 weeks
  RNA sequencing of vaginal swab samples will be performed. The RNA sequencing will measure quantities of microbes.
Change in vaginal exam findings (diameter) | From baseline to 12 weeks
  Vaginal diameter will be assessed using vaginal dilators ranging in size from small, medium, and large.
Change in vaginal exam findings (length) | From baseline to 12 weeks
  Vaginal length will be determined by measuring from vaginal cuff, apex, or cervix to posterior fourchette (mark will be made on dilator in the vagina and then measured when dilator is removed). If a dilator cannot be placed, a cotton swab will be placed into the vagina due to stenosis or poor patient tolerance and measured at the level of the posterior fourchette.
Change in sexual function | From baseline to 12 weeks
  Sexual function will be measured using the Female Sexual Functioning Index (FSFI).The FSFI is a 19-item self -reported instrument that has been previously validated to measure sexual functioning in women in clinical trials. It measures six domains of sexual functioning including arousal, orgasm, satisfaction and pain. Overall test-retest reliability coefficients are high for each domain, and the internal consistency is high with a Cronbach's alpha of 0.82 and higher. The total maximum score is 36 with a higher score indicating better functioning.
Change in Vulvovaginal symptoms (Vaginal Assessment Scale) | From baseline to 12 weeks
  The Vaginal Assessment Scale (VAS) is a recently validated clinical measurement tools to identify vulvovaginal symptoms. Patients are asked about specific symptoms over the past 4 weeks including vaginal dryness, soreness, irritation, and dyspareunia and are asked to rate them as mild, moderate, or severe. Each item is scored from 0 (none) to 3 (severe) and a composite score is calculated by taking the mean score of the items. A lower score indicates better function.
Change in Vulvovaginal symptoms (Vulvar Assessment Scale) | From baseline to 12 weeks
  The Vulvar Assessment Scale (VuAS) is a recently validated clinical measurement tools to identify vulvovaginal symptoms. Patients are asked about specific symptoms over the past 4 weeks including vaginal dryness, soreness, irritation, and dyspareunia and are asked to rate them as mild, moderate, or severe. Each item is scored from 0 (none) to 3 (severe) and a composite score is calculated by taking the mean score of the items. A lower score indicates better function.
Change in Sexual Distress | From baseline to 12 weeks
  Sexual distress will be measured using the Female Sexual Distress Scale Revised (FSDS-R), which has been shown to effectively measure sexually related personal distress in women. Higher scores indicate more distress. The revised version with 13 items was used in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Allison M Quick, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu